CLINICAL TRIAL: NCT06567717
Title: Feasibility of a Decentralized Double-Blind Randomized Controlled Trial of Zinc and Nicotinamide Riboside for the Treatment of Idiopathic Pulmonary Fibrosis
Brief Title: Zinc and Nicotinamide Riboside for Idiopathic Pulmonary Fibrosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Tanzira Zaman, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Zn-NR-001
Record Dates: First submitted 2024-08-19; First posted 2024-08-23 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: ipf; pulmonary fibrosis; idiopathic pulmonary fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Idiopathic Interstitial Pneumonias; Pulmonary Fibrosis | interventions — Zinc; nicotinamide-beta-riboside

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combination Supplements (Experimental): Zinc and nicotinamide riboside
  Interventions: Drug: Zinc; Drug: Nicotinamide riboside
- Placebo (Placebo Comparator): Placebo-controls for both zinc and nicotinamide riboside
  Interventions: Other: Placebos for zinc and nicotinamide riboside

INTERVENTIONS:
Drug: Zinc — Zinc has not previously been investigated in the treatment of IPF.
  Arms: Combination Supplements
Other: Placebos for zinc and nicotinamide riboside — These will be identical in appearance to the active substances
  Arms: Placebo
Drug: Nicotinamide riboside — Nicotinamide riboside has not previously been investigated in the treatment of IPF.
  Arms: Combination Supplements

SUMMARY:
The goal of this clinical trial is to learn if a clinical trial for idiopathic pulmonary fibrosis (IPF) can recruit and retain participants from their home to study whether a combination of zinc and nicotinamide riboside can treat iIPF. The main questions are:

Can the investigators recruit participants, and can participants complete study procedures without physically coming into specific clinical trial sites? Can people with IPF experience improvement in symptoms, quality of life, or functioning if they are take these supplements? The investigators will compare zinc and nicotinamide riboside to matched placebos (look-alike substances that contain no drug) to see if these supplements treat symptoms or lung function in people with IPF.

Participants will:

Take drug these supplements twice a day for 24 weeks. Complete pulmonary function testing and six minute walk tests with their own pulmonologists every 12 weeks. Complete a high resolution CT scan at the start and end of the study. Complete video study visits with the research team every 4 weeks. Complete surveys about their symptoms and the number of times they take the medication.

DETAILED DESCRIPTION:
This trial aims to determine the feasibility of conducting a decentralized randomized controlled trial of zinc and nicotinamide riboside versus matched placebos in addition to standard of care therapy for idiopathic pulmonary fibrosis. The investigators hypothesize that it will be feasible to remotely recruit 60 participants over 52 weeks and retain them in such a trial over 24 weeks of treatment. The investigators also hypothesize that participants will be able to complete study procedures at their local clinical facilities per standard of care without coordination by local study personnel.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Be under active treatment for IPF by a local pulmonologist
4. Age > 50 years
5. Confident diagnosis of IPF per the latest ATS/ERS/JRS/ALAT Clinical Practice Guideline on Diagnosis of IPF10

   1. Subjects must have a high-resolution computed tomography (HRCT) completed in the 6 months as part of their standard of care prior to informed consent
   2. Subjects must have HRCT pattern of definite or probable UIP
   3. Subjects without HRCT pattern of definite or probable UIP must have surgical lung biopsy as part of their standard of care showing histopathology consistent with UIP
   4. Extent of fibrotic changes must be greater than the extent of emphysema on HRCT
6. Able to take oral medication and willing to adhere to the study treatment regimen
7. Ability to utilize CS-Link, Zoom, or Doximity video conferencing for virtual study visits
8. Ability to complete PFT and 6 minute walk distance test every 12 weeks per standard of care under the order of a local treating pulmonologist
9. Ability to complete HRCT at baseline and 24 weeks per standard of care under the order of a local treating pulmonologist
10. Willingness to participate in home phlebotomy and to travel to a local Quest Diagnostics laboratory
11. Reside in one of the following states: California, Arizona, Georgia, Louisiana, Minnesota, Oregon

Exclusion Criteria:

1. FVC < 40% of predicted, DLCO < 30% of predicted, FEV1/FVC with Z-score < -1.645 or confidence interval <1.0 within 3 months of screening. If Z-scores or confidence intervals are not available, then FEV1/FVC < the lower limit of normal will be used as exclusion
2. Evidence of secondary etiologies of ILD (signs/symptoms of connective tissue disease, including ANA titer > 1:80, history of exposures related to hypersensitivity pneumonitis, history of drug related pulmonary toxicity, occupational exposures)
3. Evidence of comorbid pulmonary pathology including but not limited to asthma, tuberculosis, sarcoidosis, chronic infections
4. Any acute illness or febrile event that has not resolved at least 14 days prior to either screening or the first study visit
5. Use of tobacco-containing products within the last 3 months and/or unwillingness to abstain from use for the duration of the study
6. Participation in a clinical study involving administration of other investigational drugs in the 30 days prior to screening
7. Any condition that in the opinion of the investigators would confound the ability to interpret data from the study
8. Any comorbid condition that is likely to result in death within the next year
9. Inability to obtain reproducible, high-quality pulmonary function tests
10. Likelihood of lung transplantation in the first 12 weeks of the study
11. Use of other IPF-directed therapies beside SOC including but not limited to endothelium receptor antagonists, interferon gamma-1b, N-acetylcysteine
12. Initiation of pirfenidone or nintedanib less than 60 days prior to screening
13. Current therapy or treatment within 60 days prior to screening of any cytotoxic or immunosuppressive medications, cytokine modulating therapies within 4 weeks of the screening visit
14. Chronic prednisone usage at a dose > 10 mg daily
15. Chronic use of any restricted medications known to have significant interactions with zinc supplementation (see Section 6.5)
16. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)
17. Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
18. Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
19. History of active malignancy in the last 5 years, with the exception of carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer
20. Prior allogeneic stem cell or solid organ transplantation
21. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the participant at high risk from treatment complications

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Retention | From study activation to 78 weeks
  Feasibility is defined as 80% or more of the enrolled patients complete the 24-week treatment Additional feasibility assessments include the recruitment rate over 52 weeks and the retention rate

SECONDARY OUTCOMES:
Recruitment Rate | From study activation to 52 weeks
  Number of participants who are recruited over 52 weeks divided by 60, expressed as a percent

OTHER OUTCOMES:
Change in forced vital capacity | From enrollment to 24 weeks
  Change in the percent-predicted forced vital capacity
Change in 6 minute walk distance | From enrollment to 24 weeks
  Change in the 6 minute walk distance as expressed in meters
Change in quality of life surveys | From enrollment to 24 weeks
  Change in the score on the Living with Pulmonary Fibrosis-Symptoms and Living with Pulmonary Fibrosis-Impacts surveys
Change in diffusion capacity of the lung | From enrollment to 24 weeks
  Change in the percent-predicted diffusion capacity

CONTACTS AND LOCATIONS:
Overall Officials: Tanzira Zaman, MD, Principal Investigator — Cedars-Sinai
Locations (1):
- Cedars-Sinai, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Our study group would like to perform and publish additional analyses from the results of this trial.

REFERENCES:
- [Background] Shi B, Wang W, Korman B, Kai L, Wang Q, Wei J, Bale S, Marangoni RG, Bhattacharyya S, Miller S, Xu D, Akbarpour M, Cheresh P, Proccissi D, Gursel D, Espindola-Netto JM, Chini CCS, de Oliveira GC, Gudjonsson JE, Chini EN, Varga J. Targeting CD38-dependent NAD+ metabolism to mitigate multiple organ fibrosis. iScience. 2020 Dec 7;24(1):101902. doi: 10.1016/j.isci.2020.101902. eCollection 2021 Jan 22. PMID 33385109
- [Background] Dollerup OL, Christensen B, Svart M, Schmidt MS, Sulek K, Ringgaard S, Stodkilde-Jorgensen H, Moller N, Brenner C, Treebak JT, Jessen N. A randomized placebo-controlled clinical trial of nicotinamide riboside in obese men: safety, insulin-sensitivity, and lipid-mobilizing effects. Am J Clin Nutr. 2018 Aug 1;108(2):343-353. doi: 10.1093/ajcn/nqy132. PMID 29992272
- [Background] Conze D, Brenner C, Kruger CL. Safety and Metabolism of Long-term Administration of NIAGEN (Nicotinamide Riboside Chloride) in a Randomized, Double-Blind, Placebo-controlled Clinical Trial of Healthy Overweight Adults. Sci Rep. 2019 Jul 5;9(1):9772. doi: 10.1038/s41598-019-46120-z. PMID 31278280
- [Background] Covarrubias AJ, Perrone R, Grozio A, Verdin E. NAD+ metabolism and its roles in cellular processes during ageing. Nat Rev Mol Cell Biol. 2021 Feb;22(2):119-141. doi: 10.1038/s41580-020-00313-x. Epub 2020 Dec 22. PMID 33353981